CLINICAL TRIAL: NCT05418998
Title: Training Cognition to Improve Mobility and Listening in Older Adults with Hearing Loss: Moving from Lab to Life
Brief Title: Cognitive Training to Improve Mobility in Middle-aged and Older Adults
Acronym: HnW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Concordia University, Montreal (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Karen Li, Professor, Concordia University, Montreal
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 30011799
Record Dates: First submitted 2022-05-26; First posted 2022-06-15 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Aging; Age Related Hearing Loss
Keywords: Cognitive training; Executive function; Aging; Dual-task walking; Near-infrared spectroscopy; Hearing loss; Middle age; Mobility
MeSH Terms: conditions — Presbycusis; Hearing Loss

STUDY DESIGN:
Who Masked: Investigator
Masking Description: The investigator will be blinded to group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Executive function (EF) training (Experimental): 12 weeks of at-home EF training on a computer or iPad
  Interventions: Behavioral: Executive function (EF) training
- Wait-list control (No Intervention): This will be a comparator arm with no cognitive training. Participants will be given access to the same training program following the conclusion of the study, but no further assessment is planned.

INTERVENTIONS:
Behavioral: Executive function (EF) training — EF training will involve at-home computer- or tablet based training to improve several EF processes, including divided attention, response inhibition, switching, and working memory updating. Training session duration = 30 min x 3 session/week.
  Arms: Executive function (EF) training

SUMMARY:
The proposed study is designed to evaluate the effect of at-home executive function training on cognition and mobility in older adults with age-related hearing loss (ARHL), older adults with normal hearing, and middle-aged adults.

ELIGIBILITY:
Inclusion Criteria:

* Proficient in English (learned before age 5), can ambulate ≥ 10 meters independently, absence of cognitive impairment (neuropsychological test results in the average range compared to age norms), normal or corrected-to-normal visual acuity (ETDRS), availability of a home computer or tablet with internet connection.

Exclusion Criteria:

* Reported major depression, substance abuse or significant psychiatric disorder, uncorrected visual impairment, vestibular impairment, Parkinson's disease or other neurological disorder or sequelae, clinically significant musculoskeletal disorders, diseases affecting the ear, or damage to the ear (e.g., occupational noise), onset of hearing loss prior to adulthood.

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2020-08-30 (Actual); Primary Completion 2023-08-15 (Actual); Study Completion 2024-08-15 (Actual)

PRIMARY OUTCOMES:
Pre-training Change in auditory 2-back accuracy | baseline
  Auditory 2-back performance will be assessed under single- and dual-task conditions (i.e., while the participant is standing or simultaneously walking on a treadmill at a self-selected pace). The numbers for the task will be played through binaural speakers, and the decibel level will be individualized for each participant depending on hearing ability. Participants will be required to make a button response indicating whether the number they heard was the same or different from the number they heard two previously. Accuracy (percent correct) will be recorded. Half the participants will be given this assessment. See Outcome 5, Multi-talker, for other half.
Post-training Change in auditory 2-back accuracy | after 12 weeks
  Auditory 2-back performance will be assessed under single- and dual-task conditions (i.e., while the participant is standing or simultaneously walking on a treadmill at a self-selected pace). The numbers for the task will be played through binaural speakers, and the decibel level will be individualized for each participant depending on hearing ability. Participants will be required to make a button response indicating whether the number they heard was the same or different from the number they heard two previously. Accuracy (percent correct) will be recorded. Half the participants will be given this assessment. See Outcome 6, Multi-talker, for other half.
Pre-training Change in auditory 2-back reaction time | baseline
  Auditory 2-back performance will be assessed under single- and dual-task conditions (i.e., while the participant is standing or simultaneously walking on a treadmill at a self-selected pace). The numbers for the task will be played through binaural speakers, and the decibel level will be individualized for each participant depending on hearing ability. Participants will be required to make a button response indicating whether the number they heard was the same or different from the number they heard two previously. Reaction time (msec) will be recorded. Half the participants will be given this assessment. See Outcome 5, Multi-talker, for other half.
Post-training Change in auditory 2-back reaction time | after 12 weeks
  Auditory 2-back performance will be assessed under single- and dual-task conditions (i.e., while the participant is standing or simultaneously walking on a treadmill at a self-selected pace). The numbers for the task will be played through binaural speakers, and the decibel level will be individualized for each participant depending on hearing ability. Participants will be required to make a button response indicating whether the number they heard was the same or different from the number they heard two previously. Reaction time (msec) will be recorded. Half the participants will be given this assessment. See Outcome 6, Multi-talker, for other half.
Pre-training Multi-Talker word perception (accuracy) | baseline
  We will use the multi-talker spatial listening task for the other half of the participants, in which a presented text cue indicates which of three simultaneously presented, but spatially distributed spoken sentences to report. Traffic noise will be included to more closely simulate real- world conditions. The signal-to-noise ratio will be held constant across participants, with signal intensity set according to individual average hearing thresholds.
Post-training Multi-Talker word perception (accuracy) | after 12 weeks
  We will use the multi-talker spatial listening task for the other half of the participants, in which a presented text cue indicates which of three simultaneously presented, but spatially distributed spoken sentences to report. Traffic noise will be included to more closely simulate real- world conditions. The signal-to-noise ratio will be held constant across participants, with signal intensity set according to individual average hearing thresholds.
Pre-training Change in stride time (mean, standard deviation [SD] of stride time) | baseline
  Stride time will be assessed under single- and dual-task conditions (i.e., walking on a treadmill at a self-selected pace or while simultaneously completing the auditory 2-back task). The spatio-temporal characteristics of gait will be measured by foot pressure sensors worn on the base of the participants' shoes, with one sensor placed beneath the heel and the second sensor placed beneath the toe. The time between successive toe or heel strikes will be recorded (sec) and averaged across the trials. Those participants being assessed with Outcome 5 will perform the same walking task but in a simulated street-crossing environment.
Post-training Change in stride time (mean, standard deviation [SD] of stride time) | after 12 weeks
  Stride time will be assessed under single- and dual-task conditions (i.e., walking on a treadmill at a self-selected pace or while simultaneously completing the auditory 2-back task). The spatio-temporal characteristics of gait will be measured by foot pressure sensors worn on the base of the participants' shoes, with one sensor placed beneath the heel and the second sensor placed beneath the toe. The time between successive toe or heel strikes will be recorded (sec) and averaged across the trials. Those participants being assessed with Outcome 6 will perform the same walking task but in a simulated street-crossing environment.
Pre-training Change in stride time variability (mean, standard deviation [SD] of stride time) | baseline
  Stride time variability will be assessed under single- and dual-task conditions (i.e., walking on a treadmill at a self-selected pace or while simultaneously completing the auditory 2-back task). The spatio-temporal characteristics of gait will be measured by foot pressure sensors worn on the base of the participants' shoes, with one sensor placed beneath the heel and the second sensor placed beneath the toe. The time between successive toe or heel strikes will be recorded (sec) and the standard deviation will be taken to derive a measure of stride time variability. Those participants being assessed with Outcome 5 will perform the same walking task but in a simulated street-crossing environment.
Post-training Change in stride time variability (mean, standard deviation [SD] of stride time) | after 12 weeks
  Stride time variability will be assessed under single- and dual-task conditions (i.e., walking on a treadmill at a self-selected pace or while simultaneously completing the auditory 2-back task). The spatio-temporal characteristics of gait will be measured by foot pressure sensors worn on the base of the participants' shoes, with one sensor placed beneath the heel and the second sensor placed beneath the toe. The time between successive toe or heel strikes will be recorded (sec) and the standard deviation will be taken to derive a measure of stride time variability. Those participants being assessed with Outcome 6 will perform the same walking task but in a simulated street-crossing environment.

SECONDARY OUTCOMES:
Pre-training Montreal Cognitive Assessment (MoCA) | baseline
  Neuropsychological test to evaluate global cognitive status. Scored on 30, a score of 26 or higher is used to identify Mild Cognitive Impairment (MCI) however a score of 23 or higher is used in this study as this cut-off has been shown to lower false positivity. (Nasreddine et al., 2005)
Post-training Montreal Cognitive Assessment (MoCA) | after 12 weeks
  Neuropsychological test to evaluate global cognitive status. Scored on 30, a score of 26 or higher is used to identify Mild Cognitive Impairment (MCI) however a score of 23 or higher is used in this study as this cut-off has been shown to lower false positivity. (Nasreddine et al., 2005)
Pre-training WAIS-IV Digit Symbol Coding | baseline
  Neuropsychological test to evaluate processing speed. Subtest of the Wechsler Adult Intelligence Scale IV (WAIS; Wechsler, 2008). Scored based on correct number of symbols completed in 120 seconds.
Post-training WAIS-IV Digit Symbol Coding | after 12 weeks
  Neuropsychological test to evaluate processing speed. Subtest of the Wechsler Adult Intelligence Scale IV (WAIS; Wechsler, 2008). Scored based on correct number of symbols completed in 120 seconds.
Pre-training Trail Making Test | baseline
  Neuropsychological test to evaluate processing speed and executive functioning (Reitan, 1992). In form A, participants use a pencil to connect circles on a page in ascending numerical order. In form B, participants connect circles, alternating between ascending number and letter series. Time to complete (s) is recorded per form. Difference between Forms B and A completion times provides an index of switching, updating, and is considered a measure of executive function.
Post-training Trail Making Test | after 12 weeks
  Neuropsychological test to evaluate processing speed and executive functioning (Reitan, 1992). In form A, participants use a pencil to connect circles on a page in ascending numerical order. In form B, participants connect circles, alternating between ascending number and letter series. Time to complete (s) is recorded per form. Difference between Forms B and A completion times provides an index of switching, updating, and is considered a measure of executive function.
Pre-training D-KEFS Stroop | baseline
  Delis-Kaplan Executive Function System (D-KEFS) Color-Word Interference Test (CWIT) is a neuropsychological test to evaluate processing speed and executive functioning (adapted from Delis, Kaplan, & Kramer, 2001). A modification of the Stroop task (Stroop, 1935). In the CWIT, participants are asked to complete four conditions: colour naming, reading (both discontinued after 90 seconds), inhibition, and inhibition/switching (both discontinued after 180 seconds). Number correctly completed per condition.
Post-training D-KEFS Stroop | after 12 weeks
  Delis-Kaplan Executive Function System (D-KEFS) Color-Word Interference Test (CWIT) is a neuropsychological test to evaluate processing speed and executive functioning (adapted from Delis, Kaplan, & Kramer, 2001). A modification of the Stroop task (Stroop, 1935). In the CWIT, participants are asked to complete four conditions: colour naming, reading (both discontinued after 90 seconds), inhibition, and inhibition/switching (both discontinued after 180 seconds). Number correctly completed per condition.
Pre-training Rey Auditory Verbal Learning Test | baseline
  Neuropsychological test to evaluate verbal memory (RAVLT; Rey, A. (1941). Scored by: adding up to correctly recalled words for each trial to obtain immediate recall total; how many correctly recalled words after the 30-minute interval to obtain their delayed recall total; divided delayed recall total by the total words correctly recalled on the fifth (last) trial of the initial administration and multiplied by 100 to obtain their percentage retention value.
Post-training Rey Auditory Verbal Learning Test | after 12 weeks
  Neuropsychological test to evaluate verbal memory (RAVLT; Rey, A. (1941). Scored by: adding up to correctly recalled words for each trial to obtain immediate recall total; how many correctly recalled words after the 30-minute interval to obtain their delayed recall total; divided delayed recall total by the total words correctly recalled on the fifth (last) trial of the initial administration and multiplied by 100 to obtain their percentage retention value.
Pre-training WAIS-IV Digit span | baseline
  Neuropsychological test to evaluate short-term memory. Subtest of the Wechsler Adult Intelligence Scale IV (WAIS; Wechsler, 2008). Scored based on highest span length correctly completed.
Post-training WAIS-IV Digit span | after 12 weeks
  Neuropsychological test to evaluate short-term memory. Subtest of the Wechsler Adult Intelligence Scale IV (WAIS; Wechsler, 2008). Scored based on highest span length correctly completed.
Pre-training Subjective listening self efficacy | baseline
  Listening self-efficacy questionnaire (LSEQ: Smith, Pichora-Fuller, Watts, & La More, 2011, Int J Audiol). Asks questions about one's self-rated ability to understand conversation in a variety of contexts, without the use of hearing aids, self-rated self-efficacy (0-100%). Internal consistency (Chronbach's α) = .96 (Smith et al., 2011).
Post-training Subjective listening self efficacy | after 12 weeks
  Listening self-efficacy questionnaire (LSEQ: Smith, Pichora-Fuller, Watts, & La More, 2011, Int J Audiol). Asks questions about one's self-rated ability to understand conversation in a variety of contexts, without the use of hearing aids. Internal consistency (Chronbach's α) = .96 (Smith et al., 2011).
Pre-training Subjective balance confidence | baseline
  ABC Balance Confidence Questionnaire (Powell & Myers, 1995, J Geront: MedSci). Sixteen-item questionnaire concerning self-rated confidence (0-100%) balancing in different physical activities and contexts.
Post-training Subjective balance confidence | after 12 weeks
  ABC Balance Confidence Questionnaire (Powell & Myers, 1995, J Geront: MedSci). Sixteen-item questionnaire concerning self-rated confidence (0-100%) balancing in different physical activities and contexts.
Pre-training Mobility functioning as assessed by the Mini BESTest | baseline
  The Mini BESTest is comprised of four sub-scales to evaluate balance performance, including an anticipatory sub-scale (e.g., sit-to-stand, toe rise), a reactive postural control subscale (measures compensatory stepping when one's centre of balance is displaced in the forward, backward, or lateral position), a sensory orientation subscale (e.g., eyes closed, foam mat), and a gait subscale (e.g., walking over an obstacle).
Post-training Mobility functioning as assessed by the Mini BESTest | after 12 weeks
  The Mini BESTest is comprised of four sub-scales to evaluate balance performance, including an anticipatory sub-scale (e.g., sit-to-stand, toe rise), a reactive postural control subscale (measures compensatory stepping when one's centre of balance is displaced in the forward, backward, or lateral position), a sensory orientation subscale (e.g., eyes closed, foam mat), and a gait subscale (e.g., walking over an obstacle).
Pre-training Functional neuroimaging (fNIRS) | baseline
  Portable functional near infrared spectroscopy (BRITE MKII) will be used to assess prefrontal cortex activity during the single- and dual-task walking conditions. Sixteen detectors will be placed strategically 2.8 cm away from the optodes, eight of them will be dorsal to the optodes, while the other eight will be ventral, so that each probe has four dorsal detectors and four ventral detectors. The two probes will be placed symmetrically over the lateral prefrontal cortex and the most anterior and most ventral pair of optode-detector of each probe will be placed on Fp1/Fp2. The probes were designed based on existing configurations. Of interest are relative changes in concentration of frontal oxy-hemoglobin (HbO2: measured at absorption peak of 850nm) and deoxy-hemoglobin (HbR: measured at absorption peak of 735nm) compared to the baseline rest data.
Post-training Functional neuroimaging (fNIRS) | after 12 weeks
  Portable functional near infrared spectroscopy (BRITE MKII) will be used to assess prefrontal cortex activity during the single- and dual-task walking conditions. Sixteen detectors will be placed strategically 2.8 cm away from the optodes, eight of them will be dorsal to the optodes, while the other eight will be ventral, so that each probe has four dorsal detectors and four ventral detectors. The two probes will be placed symmetrically over the lateral prefrontal cortex and the most anterior and most ventral pair of optode-detector of each probe will be placed on Fp1/Fp2. The probes were designed based on existing configurations. Of interest are relative changes in concentration of frontal oxy-hemoglobin (HbO2: measured at absorption peak of 850nm) and deoxy-hemoglobin (HbR: measured at absorption peak of 735nm) compared to the baseline rest data.
Pre-training Standing Balance (Path length) | baseline
  Postural measures will include spatial measures (centre of pressure path length; cm) in the anterior-posterior (front and back) and medial-lateral (side-to-side) orientations.
Pre-training Standing Balance (Velocity) | baseline
  Postural measures will include temporal measures (velocity; cm/s) in the anterior-posterior (front and back) and medial-lateral (side-to-side) orientations.
Pre-training Standing Balance (Variability) | baseline
  Postural measures will include variability measures (root means square, standard deviation) in the anterior-posterior (front and back) and medial-lateral (side-to-side) orientations.
Post-training Standing Balance (Path length) | after 12 weeks
  Postural measures will include spatial measures (centre of pressure path length; cm) in the anterior-posterior (front and back) and medial-lateral (side-to-side) orientations.
Post-training Standing Balance (Velocity) | after 12 weeks
  Postural measures will include temporal measures (velocity; cm/s) in the anterior-posterior (front and back) and medial-lateral (side-to-side) orientations.
Post-training Standing Balance (Variability) | after 12 weeks
  Postural measures will include variability measures (root means square, standard deviation) in the anterior-posterior (front and back) and medial-lateral (side-to-side) orientations.

CONTACTS AND LOCATIONS:
Locations (1):
- Concordia University, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Downey R, Gagne N, Mohanathas N, Campos JL, Pichora-Fuller KM, Bherer L, Lussier M, Phillips NA, Wittich W, St-Onge N, Gagne JP, Li K. At-home computerized executive-function training to improve cognition and mobility in normal-hearing adults and older hearing aid users: a multi-centre, single-blinded randomized controlled trial. BMC Neurol. 2023 Oct 20;23(1):378. doi: 10.1186/s12883-023-03405-1. PMID 37864139